CLINICAL TRIAL: NCT02315677
Title: Nasal Intubation Using a Parker Flex-tip Endotracheal Tube With Posteriorly Facing Bevel Compared to a Nasal RAE Tube With Left Facing Bevel: A Randomized Study
Brief Title: Nasal Intubation Using a Parker Flex-tip Endotracheal Tube Compared to a Nasal RAE Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: H14-02597
Record Dates: First submitted 2014-11-24; First posted 2014-12-12 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Epistaxis
Keywords: Epistaxis; Nasal Intubation; Maxillofacial surgery
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal intubation-Standard RAE ETT (Active Comparator): This arm will receive nasal intubation with the standard RAE endotracheal tube with bevel facing left.
  Interventions: Device: Nasal Intubation with nasal RAE endotracheal tube; Device: Nasal Intubation with Parker Flex-Tip endotracheal tube
- Nasal intubation-Parker Flex-Tip ETT (Active Comparator): This arm will receive nasal intubation with the Parker Flex-tip ETT with bevel facing posteriorly.
  Interventions: Device: Nasal Intubation with nasal RAE endotracheal tube; Device: Nasal Intubation with Parker Flex-Tip endotracheal tube

INTERVENTIONS:
Device: Nasal Intubation with nasal RAE endotracheal tube — A single experienced operator with at least 5 years of clinical anesthetic experience will intubate using the standard nasal RAE endotracheal tube with bevel facing leftward.
Device: Nasal Intubation with Parker Flex-Tip endotracheal tube — A single experienced operator with at least 5 years of clinical anesthetic experience will intubate using the Parker Flex-Tip endotracheal tube with the bevel facing posteriorly.

SUMMARY:
The purpose of this study is to determine the degree of epistaxis following nasal intubation with either a nasal endotracheal (RAE) tube with bevel facing left or Parker Flex-Tip endotracheal tube with bevel facing posteriorly

The investigators hypothesize that a Parker Flex-Tip endotracheal tube when inserted with bevel facing posteriorly during nasal intubation may reduce the incidence of epistaxis intra and post-operatively. The investigators propose that using this style of endotracheal tube improves patient safety and comfort and facilitates ease and success of nasal intubation.

DETAILED DESCRIPTION:
1. Purpose

   To investigate and describe the use of a Parker Flex-Tip endotracheal tube (ETT) with a posteriorly facing bevel for nasal intubation at Vancouver Coastal Health (VCH).

   The investigators wish to demonstrate that a Parker Flex-Tip ETT with a posterior facing bevel eases ETT insertion and reduces epistaxis compared to a standard nasal RAE endotracheal tube (RAE ETT) currently used at VCH. The investigators propose that using this method improves performance and reduces complications of nasal intubation.
2. Hypothesis

   Our hypotheses are:
   * That a Parker Flex-Tip ETT with a posterior facing bevel may reduce the incidence of epistaxis
   * That a Parker Flex-Tip ETT with a posterior facing bevel may allow the anesthesiologist to successfully nasal intubate with more ease and fewer attempts.
   * That use of a Parker Flex-Tip ETT with a posterior facing bevel for nasal intubation is acceptable to anesthesiologists and patients
3. Justification

   Justification for developing a new technique Endonasal intubation is a widely performed technique that allows administration of anesthetic during oral, dental and maxillofacial surgeries while allowing unimpeded access to the surgical site. Nasal intubation poses several challenges not encountered in oropharyngeal intubation. These include advancing the endotracheal tube through the highly vascularized delicate mucosa of the nasal passage, past protruding turbinates, and maneuvering through the sharply angulated nasopharyx to access the trachea (Hall).

   The most common complication associated with endonasal intubation is epistaxis due to nasal abrasion, most commonly in the anterior part of the nasal septum, which can range from mild blood tinged mucus to massive epistaxis (Tintinalli, O'Connell, Hall). The risk of epistaxis increases with the use of excessive force, large endotracheal tube, repeated unsuccessful attempts and abnormal pharyngeal anatomy (Hall ). Rarer complications of nasal intubation include traumatic avulsion of the turbinates, turbinate fracture, retro pharyngeal laceration, and bacteremia (Williams, Hall, Dinner).

   Common techniques used to reduce the risks associated with nasal intubation include the use of vasoconstrictors in the nasal canal, lubrication of the endotracheal tube, selection of a smaller tube, mechanical dilatation of the nasal cavity, deliberate maneuvering of the tube during intubation (Hall). Other more complicated techniques have included thermosoftening and using a curved tip suction catheter to help guide the endotracheal tube (Kim, Morimoto, Wart, Seo). Overall these precautions and interventions are complicated and often ineffective in reducing complications.

   The main justification for our study is the finding from a recent study by Sugiyama . (2014) that using a Parker Flex-Tip ETT with a bent flexible tip, and advancing with the aid of an anterior flexed stylette with bevel facing posteriorly reduced the incidence of epistaxis to 4% compared to 50%, with a standard ETT. In our practice the investigators have noticed epistaxis to be present more often than not with the present nasal RAE ETT. However, the investigators have not quantified this scientifically. This significant reduction of epistaxis with a Parker Flex-Tip ETT, offers a simple and effective way to enhance patient safety and improve user ease when nasal intubation is indicated, and will improve the quality of care in our practice.

   The Parker Flex-Tip in our proposed study is identical to the Parker Flex-Tip used in the study by Sugiyama. Based on the findings by Sugiyama , the tube should allow the ETT to curve towards the oropharynx as it approaches the curve of the nasopharynx and therefore reduce impact and damage to the pharyngeal mucosa. Positioning the bevel to face posteriorly will allow the tube to slide along the posterior wall and reduce the risk of turbinate abrasion as it is advanced. The soft and curved distal tip presumably curls inward when it is advanced past the curve and a larger surface area of the tip comes into contact with the mucous membrane, reducing the pressure on the pharyngeal mucosa. Overall, the investigators predict that these modifications will increase ease of insertion and reduce the number of attempts to successful intubation, which should improve user ease and decrease risk of pharyngeal bleeding.

   The investigators aim to conduct a clinical study in 20-30 patients randomized to either the standard nasal RAE tube currently employed in our hospital or the Parker Flex-Tip ETT to demonstrate the feasibility of our technique in reducing endonasal complications at VCH.
4. Objectives - Primary and Secondary

   Our primary objective is to describe the incidence of epistaxis with the use of a Parker Flex-Tip endotracheal tube with bevel facing posteriorly during nasal intubation.

   Our secondary objectives are to describe the ease of use of a Parker Flex-Tip endotracheal tube with bevel facing posteriorly, as well as patient and operator satisfaction with the technique.
5. Research Methods

   To fulfill our objectives the investigators aim to perform a study in a clinical phase.

   A. Clinical Phase:

   The investigators plan to perform a clinical randomized study assessing the ease of use and complication rate associated with of a Parker Flex-Tip ETT with a posterior facing bevel during nasal intubation compared to a standard nasal RAE ETT.

   Study Population:

   Between 20 and 30 ASA physical status I or II patients undergoing oral or maxillofacial surgery where a nasal intubation would be appropriate for surgical anesthesia.

   ASA Physical Status 1 - A normal healthy patient

   ASA Physical Status 2 - A patient with mild systemic disease

   ASA Physical Status 3 - A patient with severe systemic disease

   ASA Physical Status 4 - A patient with severe systemic disease that is a constant threat to life

   ASA Physical Status 5 - A moribund patient who is not expected to survive without the operation.

   Patients who have documented deformities that will hinder nasal intubation, patients with a history of trauma or surgery in the area of interest, a history of epistaxis or -coagulopathies will be excluded from the study. Opioid tolerant patients taking more than 30 mg oral morphine equivalent will also be excluded from the study.

   Randomization and Blinding:

   A staff member with no clinical involvement in the study will insert the group allocation into an opaque envelope and seal the envelope. At the induction of anesthesia the envelope will be opened and the anesthesiologist will prepare the assigned tracheal tube and insert it.

   Patients will be randomly allocated to one of two groups differentiated by the type of endotracheal tube used (either a standard nasal RAE endotracheal tube with the bevel facing left or Parker Flex-Tip ET tube with bevel facing posteriorly).

   Intra operative measurements will be obtained and recorded by the attending anesthetist.

   The assessment of the presence of a post operative nose bleed or nasal pain and discomfort will be measured and recorded by an investigator who is not the attending anesthetist for the case and who is blinded to the group allocation.
6. Interventions

Patients who are scheduled for maxillofacial surgery where nasal intubation would be appropriate to deliver surgical anesthesia and who consent to participate will be studied. A single experienced operator with at least 5 years of clinical anesthetic experience will perform the clinical examination and intubation. Routine monitors will be applied and peripheral intravenous access will be established. Oxygen will be given via face mask. Anesthesia induction using intravenous fentanyl (2.5 mcg/kg), propofol (1-2 mg/kg) and rocuronium (0.5-1mg/kg) will be administered for muscle relaxation. The nostril that the patient finds easy to breathe through will be chosen for intubation. If nostril conditions are the same on both sides the right nostril will be preferred for intubation. The tracheal tube (internal diameter [ID] 7 mm for males or 6.0 mm for females) will be coated with lubricating gel and gently inserted into the patients' selected nostril. Those assigned to the Parker Flex-Tip endotracheal tube will have a curved stylette inserted in the tube before induction and the bevel will be inserted facing posteriorly. Those assigned to the standard nasal RAE endotracheal tube will have the bevel facing leftward. Both study groups will have the ETT warmed and lubricated prior to insertion.

If no resistance of the either endotracheal tube during advancement into the oropharynx is noted it will be defined as "smooth", and will be inserted into the trachea using direct laryngoscopy. In patients assigned to the Parker Flex-Tip endotracheal tube, the stylette will be withdrawn from the tube immediately after the tube passes through the nasopharynx and the tube will then be advanced into the trachea by direct laryngoscopy. If resistance is noted on insertion of either ETT it will be recorded as "impinged" and a mark will be made on the tube corresponding to the depth of insertion into the nostril to allow the distance between the tip of the tube and the mark to be measured. The assessment of the ease of insertion will only be made on the first attempt, with no manipulation applied against resistance.

The degree of epistaxis will be assessed by a blinded independent investigator immediately post intubation and up to 5 minutes post intubation, and along with ease of insertion, recorded. Quantity of epistaxis will be measured by swabbing the nasopharynx with a dry swab and measuring the difference in weight gain between the dry swab and blood soaked swab. Epistaxis will be evaluated based on the criteria established by Sugiyama . Four grades will be used:

1. No epistaxis, no blood observed on either the surface of the tube or the posterior pharyngeal wall
2. Mild epistaxis with blood apparent on the surface of the tube or posterior pharyngeal wall
3. Moderate epistaxis with pooling of blood on the posterior pharyngeal wall
4. Severe epistaxis with a large amount of blood in the pharynx impeding nasotracheal intubation and necessitating urgent orotracheal intubation

7. Study Outcome

The principal outcome is reduced epistaxis using the Parker Flex-Tip endotracheal tube when compared to the standard nasal RAE ETT with a left facing bevel.

Secondary outcomes will include:

* Ease of tube insertion
* Number of attempts to insert tube
* Post-operative patient nasal pain (Visual Analogue Score anchored at 0= no pain & 10= maximum pain) and satisfaction scores
* Operator assessment of procedure

  8. Statistical analysis

Sample size between 20 and 30. Using the results of Sugiyama (2014) study the investigators predict that the incidence of epistaxis will range between 50% and 4% in the RAE and Parker Flex-Tip group respectively. Fisher's exact test determined the sample size of at least 7 per group using α = 0.05 (two sided) and a power of 80%.

Descriptive statistics will be used to analyze success rate and to present the information gathered.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Over 16 years of age. The investigators definitely do not want to recruit anyone under age 16 yr
* Undergoing an oral or maxillofacial surgery where nasal intubation would be appropriate for surgical anesthesia
* General anesthesia and nasal intubation discussed and planned in the preoperative assessment clinic
* ASA physical status I or II patients undergoing oral or maxillofacial surgery where nasal intubation would be appropriate for surgical anesthesia.

ASA Physical Status 1 - A normal healthy patient ASA Physical Status 2 - A patient with mild systemic disease ASA Physical Status 3 - A patient with severe systemic disease ASA Physical Status 4 - A patient with severe systemic disease that is a constant threat to life ASA Physical Status 5 - A moribund patient who is not expected to survive without the operation

Exclusion Criteria:

* Patients not clinically amenable to general anesthesia
* Documented anatomical deformities in the region of interest which includes nasal passages, internal nasal turbinates and nasopharynx. These structures will henceforth be called"region of interest."
* History of trauma in the region of interest
* Previous surgery in the region of interest
* Coagulation defects
* Anticoagulant medication other than Low Dose Aspirin
* History of recurrent epistaxis
* Age less than 16 years.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reduced Epistaxis | Immediately post intubation
  The degree of epistaxis will be assessed by a blinded independent investigator immediately post intubation, and along with ease of insertion, recorded. Quantity of epistaxis will be measured by swabbing the nasopharynx with a dry swab and measuring the difference in weight gain between the dry swab and blood soaked swab. Epistaxis will be evaluated based on the criteria established by Sugiyama et al. Four grades will be used:
  1. No epistaxis, no blood observed on either the surface of the tube or the posterior pharyngeal wall
  2. Mild epistaxis with blood apparent on the surface of the tube or posterior pharyngeal wall
  3. Moderate epistaxis with pooling of blood on the posterior pharyngeal wall
  4. Severe epistaxis with a large amount of blood in the pharynx impeding nasotracheal intubation and necessitating urgent orotracheal intubation
Reduced Epistaxis | 5 minutes post intubation
  The degree of epistaxis will be assessed by a blinded independent investigator 5 minutes post intubation, and along with ease of insertion, recorded. Quantity of epistaxis will be measured by swabbing the nasopharynx with a dry swab and measuring the difference in weight gain between the dry swab and blood soaked swab. Epistaxis will be evaluated based on the criteria established by Sugiyama et al. Four grades will be used:
  1. No epistaxis, no blood observed on either the surface of the tube or the posterior pharyngeal wall
  2. Mild epistaxis with blood apparent on the surface of the tube or posterior pharyngeal wall
  3. Moderate epistaxis with pooling of blood on the posterior pharyngeal wall
  4. Severe epistaxis with a large amount of blood in the pharynx impeding nasotracheal intubation and necessitating urgent orotracheal intubation

SECONDARY OUTCOMES:
Ease of tube insertion | Immediately post intubation
  if no resistance of the either endotracheal tube during advancement into the oropharynx is noted it will be defined as "smooth", and will be inserted into the trachea using direct laryngoscopy. In patients assigned to the Parker Flex-Tip endotracheal tube, the stylette will be withdrawn from the tube immediately after the tube passes through the nasopharynx and the tube will then be advanced into the trachea by direct laryngoscopy. If resistance is noted on insertion of either ETT it will be recorded as "impinged" and a mark will be made on the tube corresponding to the depth of insertion into the nostril to allow the distance between the tip of the tube and the mark to be measured. The assessment of the ease of insertion will only be made on the first attempt, with no manipulation applied against resistance.
Number of attempts to insert tube | Immediately post intubation
Post-operative patient nasal pain | Within 2 hours after extubation
  Post-operative patient nasal pain (Visual Analogue Score anchored at 0= no pain & 10= maximum pain) and satisfaction scores. Patients will be monitored for epistaxis immediately post intubation and for up to two hours in the recovery or until patient is deemed suitable for transfer to the ward. No further monitoring required for study purposes thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Himat Vaghadia, MBBS, Principal Investigator — Vancouver Coastal Health
Locations (1):
- University of British Columbia Department of Anesthesiology, Pharmacology and Therapeutics, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Morimoto Y, Sugimura M, Hirose Y, Taki K, Niwa H. Nasotracheal intubation under curve-tipped suction catheter guidance reduces epistaxis. Can J Anaesth. 2006 Mar;53(3):295-8. doi: 10.1007/BF03022218. PMID 16527796
- [Background] Chin KJ, Perlas A. Ultrasonography of the lumbar spine for neuraxial and lumbar plexus blocks. Curr Opin Anaesthesiol. 2011 Oct;24(5):567-72. doi: 10.1097/ACO.0b013e32834aa234. PMID 21822134
- [Background] Hall CE, Shutt LE. Nasotracheal intubation for head and neck surgery. Anaesthesia. 2003 Mar;58(3):249-56. doi: 10.1046/j.1365-2044.2003.03034.x. PMID 12603455
- [Background] Williams AR, Burt N, Warren T. Accidental middle turbinectomy: a complication of nasal intubation. Anesthesiology. 1999 Jun;90(6):1782-4. doi: 10.1097/00000542-199906000-00039. No abstract available. PMID 10360881
- [Background] Dost P, Armbruster W. Nasal turbinate dislocation caused by nasotracheal intubation. Acta Anaesthesiol Scand. 1997 Jun;41(6):795-6. doi: 10.1111/j.1399-6576.1997.tb04787.x. PMID 9241346
- [Background] Tintinalli JE, Claffey J. Complications of nasotracheal intubation. Ann Emerg Med. 1981 Mar;10(3):142-4. doi: 10.1016/s0196-0644(81)80379-4. PMID 7469154
- [Background] Dinner M, Tjeuw M, Artusio JF Jr. Bacteremia as a complication of nasotracheal intubation. Anesth Analg. 1987 May;66(5):460-2. doi: 10.1213/00000539-198705000-00017. No abstract available. PMID 3578854
- [Background] O'Connell JE, Stevenson DS, Stokes MA. Pathological changes associated with short-term nasal intubation. Anaesthesia. 1996 Apr;51(4):347-50. doi: 10.1111/j.1365-2044.1996.tb07746.x. PMID 8686823
- [Background] Sugiyama K, Manabe Y, Kohjitani A. A styletted tracheal tube with a posterior-facing bevel reduces epistaxis during nasal intubation: a randomized trial. Can J Anaesth. 2014 May;61(5):417-22. doi: 10.1007/s12630-014-0156-3. Epub 2014 Mar 28. PMID 24740408
- [Background] Seo KS, Kim JH, Yang SM, Kim HJ, Bahk JH, Yum KW. A new technique to reduce epistaxis and enhance navigability during nasotracheal intubation. Anesth Analg. 2007 Nov;105(5):1420-4, table of contents. doi: 10.1213/01.ane.0000281156.64133.bd. PMID 17959976
- [Background] Watt S, Pickhardt D, Lerman J, Armstrong J, Creighton PR, Feldman L. Telescoping tracheal tubes into catheters minimizes epistaxis during nasotracheal intubation in children. Anesthesiology. 2007 Feb;106(2):238-42. doi: 10.1097/00000542-200702000-00010. PMID 17264716
- [Background] Kim YC, Lee SH, Noh GJ, Cho SY, Yeom JH, Shin WJ, Lee DH, Ryu JS, Park YS, Cha KJ, Lee SC. Thermosoftening treatment of the nasotracheal tube before intubation can reduce epistaxis and nasal damage. Anesth Analg. 2000 Sep;91(3):698-701. doi: 10.1097/00000539-200009000-00038. PMID 10960403
- [Derived] Earle R, Shanahan E, Vaghadia H, Sawka A, Tang R. Epistaxis during nasotracheal intubation: a randomized trial of the Parker Flex-Tip nasal endotracheal tube with a posterior facing bevel versus a standard nasal RAE endotracheal tube. Can J Anaesth. 2017 Apr;64(4):370-375. doi: 10.1007/s12630-017-0813-4. Epub 2017 Jan 11. PMID 28078544